CLINICAL TRIAL: NCT01519206
Title: Evaluation of the Efficacy and Safety of the Ulthera® System for Lifting and Tightening of the Face and Neck Following an Increased Density Treatment.
Brief Title: Lifting and Tightening of the Face and Neck Following an Increased Density Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ULT-124
Record Dates: First submitted 2011-12-08; First posted 2012-01-26 (Estimated); Results first posted 2014-06-02 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Skin Laxity
Keywords: Ulthera® System; Ultherapy™ Treatment; Ulthera, Inc.
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultherapy treatment (Experimental): Ulthera System Treatment
  Interventions: Device: Ulthera System Treatment

INTERVENTIONS:
Device: Ulthera System Treatment — Focused ultrasound energy delivered below the surface of the skin.
  Other Names: Ultherapy™; Ulthera, Inc.; Ultrasound treatment for skin tightening

SUMMARY:
The purpose of this study is to evaluate the Ulthera® System for obtaining lift and tightening of the cheek tissue, reduction of jowling, and improving jawline definition and/or submental skin laxity when increased density treatment is applied.

DETAILED DESCRIPTION:
All enrolled study subjects will receive one full face and neck Ultherapy™ treatment. Pre- and post-treatment photos will be taken. Subjects will be required to return for follow-up visits at 60 days, 90 days, 180 days and 1 year following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 30 to 65 years
* Subject in good health
* Desires lift and tightening of cheek tissue, reduction of jowling, improvement of jawline definition and/or submental skin laxity
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the followup period
* Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study

Exclusion Criteria:

* Presence of an active systemic or local skin disease that may affect wound healing
* Severe solar elastosis
* Excessive subcutaneous fat on the cheeks
* Excessive skin laxity on the lower face and neck
* Significant scarring in areas to be treated
* Significant open facial wounds or lesions
* Severe or cystic acne on the face
* Presence of a metal stent or implant in the facial area to be treated, a pacemaker, or cochlear implants

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-08; Primary Completion 2012-02 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy Geronemus, M.D., Principal Investigator — Laser & Skin Surgery Center of NY
Locations (1):
- Laser & Skin Surgery Center of NY, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-five (35) subjects were enrolled, 3 were deemed screen failures. Thirty-two (32) received study treatment. The first subject was treated on August 3, 2011 and the last subject was treated on 11/28/2011. The last patient follow-up for the trial was 11/21/2012.
Groups:
- Ultherapy Treatment: Study subjects received a full face Ultherapy treatment delivering approximately 500 treatment lines at two treatment depths, i.e., 4.5mm and 3.0mm depth.
Period: Overall Study
Arm/Group | Ultherapy Treatment
Started | 32
Completed | 27
Not Completed | 5
Not completed — Lost to Follow-up | 3
Not completed — Missed Visit | 2

BASELINE CHARACTERISTICS:
Arm/Group | Ultherapy Treatment
Number analyzed (Participants) | 32
Age, Continuous [Mean (Full Range); unit: years] | 55 [44 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 30
  African American/Black | 1
  Hispanic/Latino | 1
Region of Enrollment [Number; unit: participants]
  United States | 32
Fitzpatrick Skin Type [Number; unit: participants] — Skin Type I = White; very fair, red or blonde hair blue eyes; freckles; Always burns, never tans Skin Type II = White, fair, red or blond hair; blue, hazel or green eyes; Usually burns, tans with difficulty Skin Type III = Cream white; fair with any eye or hair color (common); Sometimes mild burn, gradually tans Skin Type IV = Brown; typical Mediterranean Caucasian skin; Rarely burns, tans with ease Skin Type V = Dark Brown; mid-eastern skin types; Very rarely burns, tans easily Skin Type VI = Black; Never burns, tans very easily
  participants
    I | 1
    II | 24
    III | 6
    IV | 0
    V | 1
    VI | 0
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m˄2] | 23.3 [18.0 to 30.2]

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Overall Lifting and Tightening of Skin
Description: Improvement in overall lifting and tightening of skin was completed by three masked assessors, completing a qualitative assessment of pre- and post-treatment photographs. Masked photo pairs of pre/post treatment photos of each treated subject were provided to each assessor. Each photo pair was consistent in lighting, position, focus. The visit interval of each photo was NOT marked. Each assessor's review was completed independently, with no input from others, assessing the photos for improvement. If improvement was seen, the blinded assessor was to choose the post-treatment photo. Categories of assessment included Improved, No Change, or Incorrect post-treatment photo chosen. The majority assessment among the 3 blinded assessors for each subject was reported.
Time Frame: Baseline to 90 days post treatment
Population: Thirty-five (35) subjects were enrolled; 3 were screen failures. Thirty-two (32) subjects received study treatment. Three (3) subjects were lost-to-follow-up.
Measure: Number; unit: percentage of participants improved
Arm/Group | Ultherapy Treatment
Number analyzed (Participants) | 29
percentage of participants improved | 48

2. Secondary Outcome: Overall Aesthetic Improvement at 60 Days, 90 Days, 180 Days and 1 Year Post-treatment.
Description: Improvement was assessed based on Global Aesthetic Improvement Scale (GAIS) scores. The GAIS was completed based on a live assessment of the subject and a photographic assessment comparing post-treatment photos to baseline photos. The PGAIS was completed by a clinician assessor; SGAIS was completed by the study subject. The GAIS is a 5-point scale (1-5) describing an overall assessment as follows:
  1. - Very Much Improved
  2. - Much Improved
  3. - Improved
  4. - No Change
  5. - Worse
Time Frame: Baseline to 60 days, 90 days, 180 days and 1 year post-treatment
Population: Three (3) subjects were lost-to-follow-up. Two (2) additional subjects missed the 1 year visit.
Measure: Number; unit: Percentage of Participants
Groups:
- Treated Subjects GAIS Data - 60 Days Post-treatment; Treated Subjects GAIS Data - 90 Days Post-treatment; Treated Subjects GAIS Data - 180 Days Post-treatment; Treated Subjects GAIS Data - 1 Year Post-treatment: Study subjects received a full face Ultherapy treatment delivering approximately 500 treatment lines at two treatment depths, i.e., 4.5mm and 3.0mm depth.
Arm/Group | Treated Subjects GAIS Data - 60 Days Post-treatment | Treated Subjects GAIS Data - 90 Days Post-treatment | Treated Subjects GAIS Data - 180 Days Post-treatment | Treated Subjects GAIS Data - 1 Year Post-treatment
Number analyzed (Participants) | 29 | 29 | 29 | 27
Percentage of Participants
  PGAIS - Very Much Improved | 7 | 14 | 7 | 7
  PGAIS - Much Improved | 28 | 24 | 10 | 22
  PGAIS - Improved | 59 | 41 | 48 | 70
  PGAIS - No Change | 7 | 21 | 31 | 0
  PGAIS - Worse | 0 | 0 | 3 | 0
  SGAIS - Very Much Improved | 3 | 3 | 0 | 4
  SGAIS - Much Improved | 10 | 17 | 17 | 7
  SGAIS - Improved | 48 | 41 | 52 | 41
  SGAIS - No Change | 34 | 34 | 24 | 41
  SGAIS - Worse | 3 | 3 | 7 | 7

3. Secondary Outcome: Subjects' Assessment of Pain
Description: Subjects' sensory response to the Ulthera treatment exposures were recorded for each anatomical region treated using a validated Numeric Rating Scale (0-10), with 1 representing no pain and 10 representing the worst pain possible. Subjects rated pain for each transducer, in each treatment region. For statistical analyses, NRS scores were averaged for each transducer depth.
Time Frame: During Ulthera treatment
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Ultherapy Treatment
Number analyzed (Participants) | 32
Units on a scale
  4.5mm Transducer | 4.6 [0 to 9]
  3.0mm Transducer | 3.6 [0 to 7]

4. Secondary Outcome: Subject Satisfaction at 90 Days, 180 Days and 1 Year Post-treatment
Description: Subject satisfaction was determined by scores on a patient satisfaction questionnaire (PSQ) completed at 90 days, 180 days and 1 year post-treatment. Subjects indicated how satisfied they were with their study treatment, i.e., Very Satisfied, Satisfied, Dissatisfied, Very Dissatisfied. Pre-treatment and post-treatment photographs were available for viewing at each follow-up visit interval. Subjects also had a mirror available for real time assessment, comparing their image in the mirror with pre-treatment and post-treatment photos.
Time Frame: Baseline to 90 days, 180 days and 1 year post-treatment
Population: Three (3) subjects were lost-to-follow-up. Two (2) subjects missed the 1 year visit.
Measure: Number; unit: Percentage of Participants
Groups:
- Treated Subjects PSQ Data - 90 Days Post-treatment; Treated Subjects PSQ Data - 180 Days Post-treatment; Treated Subjects PSQ Data - 1 Year Post-treatment: Study subjects received a full face Ultherapy treatment delivering approximately 500 treatment lines at two treatment depths, i.e., 4.5mm and 3.0mm depth.
Arm/Group | Treated Subjects PSQ Data - 90 Days Post-treatment | Treated Subjects PSQ Data - 180 Days Post-treatment | Treated Subjects PSQ Data - 1 Year Post-treatment
Number analyzed (Participants) | 29 | 29 | 27
Percentage of Participants
  Very Satisfied | 21 | 10 | 7
  Satisfied | 48 | 59 | 41
  Dissatisfied | 24 | 21 | 37
  Very Dissatisfied | 7 | 10 | 15

ADVERSE EVENTS:
Time Frame: Adverse events were assessed during the entire study period, i.e., 1 year post-treatment.
Arm/Group | Ultherapy Treatment
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

LIMITATIONS AND CAVEATS:
3-D digital imaging was not completed, thus quantitative measure of submental skin lift was not obtained.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No